CLINICAL TRIAL: NCT00692510
Title: A Phase I, Double Blind, Randomized, Two-Way Cross Over, Single- Centre Study in Healthy CYP2D6 Extensive Metabolizers and Poor Metabolizers to Investigate the Potential of AZD3480 to Inhibit Cytochrome P450 1A2, 2C19, 3A4, 2C8, 2B6 and UGT1A1 Activity
Brief Title: Drug Interaction Study Between AZD3480 and Cytochrome P450
Acronym: Cocktail
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans-Göran Hårdemark, MD, PhD, Medical Science Director, AstraZeneca R&D Södertälje, Sweden
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D3690C00016; EudraCt nr 2007-002456-10
Record Dates: First submitted 2008-05-29; First posted 2008-06-06 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Metabolism; Alzheimer's Disease
Keywords: AZD3480; Cocktail; caffeine; bupropion; omeprazole; midazolam; rosiglitazone; metabolism; Drug Drug Interaction
MeSH Terms: conditions — Alzheimer Disease | interventions — ispronicline; Caffeine; Bupropion; Rosiglitazone; Omeprazole; Midazolam; Bilirubin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD3480 + cocktail
  Interventions: Drug: AZD3480; Drug: Cocktail mix (Caffeine, Bupropion, Rosiglitazone, Omeprazole, Midazolam, Bilirubin)
- 2 (Placebo Comparator): Placebo + cocktail
  Interventions: Drug: Placebo; Drug: Cocktail mix (Caffeine, Bupropion, Rosiglitazone, Omeprazole, Midazolam, Bilirubin)

INTERVENTIONS:
Drug: AZD3480 — Capsule, oral, dose once daily, 7 days
  Arms: 1
Drug: Placebo — Capsule, oral, dose once daily, 7 days
  Arms: 2
Drug: Cocktail mix (Caffeine, Bupropion, Rosiglitazone, Omeprazole, Midazolam, Bilirubin) — Cocktail mix which contains the following:
  CYP1A2 (Caffeine), CYP2B6 (Bupropion), CYP2C8 (Rosiglitazone), CYP2C19 (Omeprazole), CYP3A4 (Midazolam), UGT1A1 (Bilirubin)
  single dose of mix

SUMMARY:
The purpose of the study is to evaluate if AZD3480 inhibits Cytochrome P450 1A2, 2C19, 3A4, 2C8, 2B6 and UGT1A1 activity.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent
* Clinically normal physical findings and laboratory values

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma within three weeks before the first dose
* History of clinically significant disease
* Use of prescribed medication during the 2 weeks before administration of the first dose of investigational product

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during the treatment periods

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Göran Hårdemark, MD, Study Director — AstraZeneca R&D, Södertälje, Sweden; Cyril Clarke, MD, Principal Investigator — ICON Development Solutions Manchester, Manchester Science Park, Manchester, UK
Locations (1):
- Research Site, Uppsala, Sweden